CLINICAL TRIAL: NCT06452524
Title: The Precondition of Retinopathy of Prematurity on Visual Acuity, Refraction, Biometric Values, Retinal and Choroidal Thickness in School-Aged Children
Brief Title: Prematurity and Ophthalmological Changes
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ali Kutay KILINÇ, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: AKU749K
Record Dates: First submitted 2024-05-24; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Retinopathy of Prematurity; Myopia
Keywords: Biometry; foveal thickness; choroidal thickness; laser photocoagulation; OCT; prematurity; retinopathy of prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Myopia; Premature Birth | interventions — Tomography, Optical Coherence; Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ROP-Tx Group: less than 37 weeks were divided into three groups: 29 children born prematurely who were treated with laser photocoagulation
  Interventions: Device: axial length (AU) and anterior chamber depth (ACD), optical coherence tomography (OCT)
- ROP-non-Tx Group: 26 children who developed ROP and did not need treatment
  Interventions: Device: axial length (AU) and anterior chamber depth (ACD), optical coherence tomography (OCT)
- Premature Group: 25 children who did not develop ROP
  Interventions: Device: axial length (AU) and anterior chamber depth (ACD), optical coherence tomography (OCT)
- Control Group: 27 healthy children with a history of full-term born
  Interventions: Device: axial length (AU) and anterior chamber depth (ACD), optical coherence tomography (OCT)

INTERVENTIONS:
Device: axial length (AU) and anterior chamber depth (ACD), optical coherence tomography (OCT) — Non-cycloplegic and cycloplegic refraction, best corrected visual acuity (BCVA), axial length (AU) and anterior chamber depth (ACD), optical coherence tomography (OCT) macular and OCT subfoveal choroidal measurements were performed in all cases.
  Other Names: ROP-Tx Group; ROP-non-Tx Group; Premature Group; Control Group

SUMMARY:
Ophthalmological differences in school-aged children with and without a history of retinopathy of prematurity

DETAILED DESCRIPTION:
Aims: To compare functional (visual acuity and refractive error) and anatomical (biometric values, foveal and choroidal thickness) ophthalmological differences in school-aged children with and without a history of retinopathy of prematurity (ROP).

Settings and Design: Prospective Cross-Sectional Study

Methods and Material: The study was conducted prospectively in the ophthalmology department of Ankara Bilkent City Hospital. Subjects were divided into three groups: 29 children who were treated with laser photocoagulation (ROP-TxGroup), 26 children who developed ROP and did not need treatment (ROP-non-TxGroup), and 25 children who did not develop ROP (Premature Group). The 27 healthy children with a history of full-term born (Control Group), who were in a similar age group for 'control eye examination', were accepted as the control group. A total of 107 patients and 211 eyes were included in the study. Non-cycloplegic and cycloplegic refraction, best corrected visual acuity (BCVA), keratometry, axial length (AL) and anterior chamber depth (ACD), optical coherence tomography (OCT) macular and OCT subfoveal choroidal measurements were performed in all cases.

ELIGIBILITY:
Inclusion Criteria:

Children with a history of ROP

Exclusion Criteria:

Stage 4-5 ROP, Presence of media opacities (such as cataract) Ocular trauma or ocular surgery Hydrocephalus or grade 3 and above intracerebral hemorrhage, Uncooperative children

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The files of babies born between 2008 and 2016 and taken for ROP scan in the ophthalmology department were randomly separated by archive scanning. International Classification of Retinopathy of Prematurity (ICROP) was used as classification criteria. Although ICROP was used as screening criteria, every patient suspected by the paediatrician was examined. When the children of the volunteer families reached the age of 5-13, their children were called for examination.
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Spherical Equivalents | 4mounth after the procedure
  Dioptre
K1 Flat and K2 Steep | 4mounth after the procedure
  Dioptre
Axial Length | 4mounth after the procedure
  Milimeter
Anterior Chamber Depth | 4mounth after the procedure
  Milimeter
Astigmatism | 4mounth after the procedure
  Dioptre
Best Corrected Visual Acuity | 4mounth after the procedure
  logMAR
Macular and Choroidal Thickness | 4mounth after the procedure
  Micrometer

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kutay KILINÇ, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided